CLINICAL TRIAL: NCT04483778
Title: Phase I Study of B7H3 CAR T Cell Immunotherapy for Recurrent/Refractory Solid Tumors in Children and Young Adults
Brief Title: B7H3 CAR T Cell Immunotherapy for Recurrent/Refractory Solid Tumors in Children and Young Adults
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Seattle Children's Hospital (Other)
Responsible Party: Principal Investigator, Colleen Annesley, Medical Director, Seattle Children's Therapeutics, Seattle Children's Hospital
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: STRIvE-02
Record Dates: First submitted 2020-07-14; First posted 2020-07-23 (Actual); Last update posted 2025-11-20 (Actual); Status verified 2025-11

CONDITIONS: Pediatric Solid Tumor; Germ Cell Tumor; Retinoblastoma; Hepatoblastoma; Wilms Tumor; Rhabdoid Tumor; Carcinoma; Osteosarcoma; Ewing Sarcoma; Rhabdomyosarcoma; Synovial Sarcoma; Clear Cell Sarcoma; Malignant Peripheral Nerve Sheath Tumors; Desmoplastic Small Round Cell Tumor; Soft Tissue Sarcoma; Neuroblastoma; Melanoma
Keywords: CAR T cell; Pediatric; Young adults; Non-CNS solid tumor
MeSH Terms: conditions — Neoplasms, Germ Cell and Embryonal; Retinoblastoma; Hepatoblastoma; Wilms Tumor; Rhabdoid Tumor; Carcinoma; Osteosarcoma; Sarcoma, Ewing; Rhabdomyosarcoma; Sarcoma, Synovial; Sarcoma, Clear Cell; Neurofibrosarcoma; Desmoplastic Small Round Cell Tumor; Sarcoma; Neuroblastoma; Melanoma | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- SCRI-CARB7H3(s) (Experimental): Autologous CD4+ and CD8+ T-cells genetically modified to express an B7H3-specific CAR
  Interventions: Biological: second generation 4-1BBζ B7H3-EGFRt-DHFR
- SCRI-CARB7H3(s)x19 (Experimental): Autologous CD4+ and CD8+ T-cells genetically modified to a bispecific B7H3xCD19 CAR
  Interventions: Biological: second generation 4-1BBζ B7H3-EGFRt-DHFR(selected) and a second generation 4-1BBζ CD19-Her2tG
- SCRI-CARB7H3(s)x19 plus pembrolizumab (Experimental): Autologous CD4+ and CD8+ T-cells genetically modified to express a bispecific B7H3xCD19 CAR given in combination with pembrolizumab
  Interventions: Biological: second generation 4-1BBζ B7H3-EGFRt-DHFR(selected) and a second generation 4-1BBζ CD19-Her2tG; Drug: Pembrolizumab

INTERVENTIONS:
Biological: second generation 4-1BBζ B7H3-EGFRt-DHFR — Autologous CD4+ and CD8+ T-cells lentivirally transduced to express a second generation 4-1BBζ B7H3-EGFRt-DHFR
  Arms: SCRI-CARB7H3(s)
Biological: second generation 4-1BBζ B7H3-EGFRt-DHFR(selected) and a second generation 4-1BBζ CD19-Her2tG — Autologous CD4+ and CD8+ T-cells lentivirally transduced to express a second generation 4-1BBζ B7H3-EGFRt-DHFR(selected) and a second generation 4-1BBζ CD19-Her2tG
  Arms: SCRI-CARB7H3(s)x19; SCRI-CARB7H3(s)x19 plus pembrolizumab
Drug: Pembrolizumab — SCRI-CARB7H3(s)x19 plus pembrolizumab
  Arms: SCRI-CARB7H3(s)x19 plus pembrolizumab

SUMMARY:
This is a phase I, open-label, non-randomized study that will enroll pediatric and young adult research participants with relapsed or refractory non-CNS solid tumors to evaluate the safety, feasibility, and efficacy of administering T cell products derived from the research participant's blood that have been genetically modified to express a B7H3-specific receptor (chimeric antigen receptor, or CAR) that will target and kill solid tumors that express B7H3. On Arm A of the study, research participants will receive B7H3-specific CAR T cells only. On Arm B of the study, research participants will receive CAR T cells directed at B7H3 and CD19, a marker on the surface of B lymphocytes, following the hypothesis that CD19+ B cells serving in their normal role as antigen presenting cells to T cells will promote the expansion and persistence of the CAR T cells. Arm A CAR T cells include the protein EGFRt and Arm B CAR T cells include the protein HER2tG. These proteins can be used to both track and destroy the CAR T cells in case of undue toxicity. The primary objectives of the study will be to determine the feasibility of manufacturing the cell products, the safety of the T cell product infusion, to determine the maximum tolerated dose of the CAR T cells products, to describe the full toxicity profile of each product, and determine the persistence of the modified cell in the participant's body on each arm. Participants will receive a single dose of T cells comprised of two different subtypes of T cells (CD4 and CD8 T cells) felt to benefit one another once administered to the research participants for improved potential therapeutic effect. The secondary objectives of this protocol are to study the number of modified cells in the patients and the duration they continue to be at detectable levels. The investigators will also quantitate anti-tumor efficacy on each arm. Participants who experience significant and potentially life-threatening toxicities (other than clinically manageable toxicities related to T cells working, called cytokine release syndrome) will receive infusions of cetuximab (an antibody commercially available that targets EGFRt) or trastuzumab (an antibody commercially available that targets HER2tG) to assess the ability of the EGFRt on the T cells to be an effective suicide mechanism for the elimination of the transferred T cell products.

ELIGIBILITY:
Inclusion Criteria:

* Participants age ≤ 26 years at the time of consent for study participation; the first 2 participants enrolled and treated with CAR T cells in both Arms A and B will be ≥ 15 years. and ≤ 26 years at time of consent for study participation
* Histologically diagnosed malignant, non-primary CNS solid tumor
* Evidence of refractory or recurrent disease
* Lansky or Karnofsky score ≥ 50
* Life expectancy ≥ 8 weeks
* Recovered from significant acute toxic effects of all prior chemotherapy, immunotherapy and radiotherapy
* If no apheresis product or usable T cell product is available, all chemotherapy has been discontinued ≥ 7 days prior to enrollment
* If no apheresis or usable T cell product is available, all biologic therapy has been discontinued ≥ 7 days prior to enrollment
* If no apheresis product or T cell product is available, all systemic corticosteroid therapy has been discontinued ≥ 7 days prior to enrollment (physiologic replacement dosing is allowed)
* If no apheresis product or usable T cell product is available, at least 3 half-lives or 30 days (whichever is shorter) from time of last dose of anti-tumor directed antibody therapy (including checkpoint inhibitor) at time of enrollment
* If no apheresis product or usable T cell product is available, at least 6 weeks post last dose of myeloablative therapy and autologous and/or allogeneic stem cell transplant, or non-myeloablative therapy and allogeneic stem cell transplant (all timed from stem cell infusion). Participants who receive autologous stem cell infusion following non-myeloablative therapy are eligible once all other eligibility requirements are met.
* If no apheresis product or usable T cell product is available, participants who have received genetically modified cell therapy must be at least 30 days from most recent cell infusion prior to enrollment
* If no apheresis product or usable T cell product is available, participants with neuroblastoma must be at least 12 weeks from I131 MIBG therapy.
* Adequate organ function
* Adequate laboratory values
* Participant is able to tolerate apheresis (including placement of temporary apheresis catheter, if necessary), or already has an apheresis product available for use in manufacturing.
* Participants of childbearing potential must agree to use highly effective contraception

Exclusion Criteria:

* Presence of active malignancy other than primary malignant solid tumor diagnosis
* Current relevant CNS pathology
* Receiving external beam radiation therapy at time of enrollment
* Presence of active GVHD, or receiving immunosuppressive therapy for treatment or prevention of GVHD within 4 weeks prior to enrollment
* Participant is pregnant or breastfeeding
* Participant has presence of active severe infection
* Participant has presence of any condition that, in the option of an investigator, would prohibit the participant from undergoing treatment under this protocol
* Participant has primary immunodeficiency syndrome
* Unwilling or unable to provide consent/assent for participation in the study and 15 year follow up period

Ages: 0 Years to 26 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 68 (Estimated)
Dates: Start 2020-07-13 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2040-12 (Estimated)

PRIMARY OUTCOMES:
Assess the safety and tolerability of cellular immunotherapy utilizing ex-vivo expanded autologous T cells genetically modified to express B7H3-specific CAR (Arm A) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
Assess the safety and tolerability of cellular immunotherapy utilizing ex-vivo expanded autologous T cells genetically modified to express a bispecific B7H3xCD19 CAR (Arm B) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To assess the safety and tolerability of cellular immunotherapy utilizing ex-vivo expanded autologous T cells genetically modified to express a bispecific B7H3xCD19 CAR given in combination with pembrolizumab (Arm C) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized to determine maximal tolerated dose
To determine the maximum tolerated dose (MTD) of B7H3-specific CAR (Arm A) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized to determine maximal tolerated dose
To determine the maximum tolerated dose of bispecific B7H3xCD19 CAR (Arm B) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To determine the feasibility of administration of pembrolizumab in combination with bispecific B7H3xCD19 CAR (Arm C) | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To assess the dose limiting toxicities (DLTs) and describe the full toxicity profile for each study arm | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To assess the feasibility of manufacturing B7H3 specific CARs from patient-derived lymphocytes | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized
To assess the feasibility of manufacturing B7H3xCD19 bispecific CARs from patient-derived lymphocytes | 28 days
  Type, frequency, severity, and duration of adverse events will be tabulated and summarized

SECONDARY OUTCOMES:
Determine the duration of in vivo persistence of adoptively transferred T cells in the peripheral blood and compare engraftment between T cell products and treatment arms | 84 days
  Presence of CAR T cells in the peripheral blood will be assessed
Determine the magnitude of in vivo persistence of adoptively transferred T cells in the peripheral blood and compare engraftment between T cell products | 84 days
  Number of CAR T cells in the peripheral blood will be assessed
Quantitate anti-tumor responses by measuring changes in tumor burden using disease-specific evaluations | 84 days
  Presence of CAR T cells in the peripheral blood will be assessed
Describe the relative expansion and persistence of the CAR T cell product and retention of function for B7H3xCD19 bispecific CARs determined by maintenance of B cell aplasia (BCA) with and without pembrolizumab | 84 days
  Presence of CAR T cells in the peripheral blood will be assessed

OTHER OUTCOMES:
Evaluate for the presence of B7H3 CAR T cells in tumor tissue and/or normal tissue if a tissue biopsy, tumor biopsy, or resection is clinically indicated post-treatment | 84 days
  Tumor tissue, when obtained, will be assessed for the presence of adoptively transferred CAR T cells
Evaluate B7H3 antigen expression in tumor tissue and/or normal tissue if a tissue biopsy, tumor biopsy, or resection is available | 84 days
  Tumor tissue, when obtained, will be assessed for the presence of B7H3 antigen
Analyze blood, bone marrow, CSF, normal tissue, and/or tumor tissue for biomarkers of safety and/or anti-tumor activity | 84 days
  If a tissue biopsy, tumor biopsy, or resection is clinically indicated post-treatment, pathology will be assessed for the presence of B7H3 CAR T cells
Assess the efficacy of infusional cetuximab and/or trastuzumab in ablating transferred T cells and ameliorating acute toxicities in treated participants | 84 days
  Biologic specimens, when obtained, will be assessed for biomarkers of safety and/or anti-tumor efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Albert, MD, Principal Investigator — Seattle Children's Hospital
Locations (1):
- Seattle Children's Hospital, Seattle, Washington, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pinto N, Albert CM, Taylor MR, Ullom HB, Wilson AL, Huang W, Wendler J, Pattabhi S, Seidel K, Brown C, Gustafson JA, Rawlings-Rhea SD, Cheeney SHE, Burleigh K, Gustafson HH, Orentas RJ, Vitanza NA, Gardner RA, Jensen MC, Park JR. STRIvE-02: A First-in-Human Phase I Study of Systemically Administered B7-H3 Chimeric Antigen Receptor T Cells for Patients With Relapsed/Refractory Solid Tumors. J Clin Oncol. 2024 Dec 10;42(35):4163-4172. doi: 10.1200/JCO.23.02229. Epub 2024 Sep 10. PMID 39255444